CLINICAL TRIAL: NCT05871073
Title: Dexamethasone as Adjuvant to Ropivacaine in Wound Infiltration for Postoperative Analgesia Following Spinal Surgery: A Randomized, Double-Blinded, Controlled Trial
Brief Title: Dexamethasone as Adjuvant to Ropivacaine in Wound Infiltration for Postoperative Analgesia Following Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Fattouma Bourguiba (Other)
Responsible Party: Principal Investigator, Atef Ben Nsir, UNIVERSITY OF MONAASTIR, University Hospital Fattouma Bourguiba
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PAIN MANAGMENT IN SURGERY
Record Dates: First submitted 2023-04-11; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Disc Herniation; Lumbar Spondylolisthesis; Lumbar Spine Instability
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement; Spondylolisthesis | interventions — Ropivacaine; Single Person; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine 0.75% Injectable Solution (Experimental): Wound Infiltration for Postoperative Analgesia After Spinal Surgery
  Interventions: Drug: Ropivacaine 0.75% Injectable Solution
- Dexamethasone 8mg (Experimental): Wound Infiltration for Postoperative Analgesia After Spinal Surgery
  Interventions: Drug: Ropivacaine 0.75% Injectable Solution; Drug: dexamethasone 8mg

INTERVENTIONS:
Drug: Ropivacaine 0.75% Injectable Solution — WOUND INFILTRATION AFTER SPINAL SURGERY
  Other Names: Alone
Drug: dexamethasone 8mg — WOUND INFILTRATION AFTER SPINAL SURGERY
  Other Names: with Ropivacaine 0.75% Injectable Solution
  Arms: Dexamethasone 8mg

SUMMARY:
Introduction: Improving postoperative pain management after spinal surgery is a significant challenge for surgeons and anesthesiologists. Pain following spinal surgery, can lead to significant morbidity, limit early mobility, and increase the risk of chronic pain. This trial examines the analgesic effects of dexamethasone as an adjuvant to ropivacaine in wound infiltration after lumbar surgery.

Methods: In this study, we randomly assigned sixty patients undergoing lumbar laminectomy and/or osteosynthesis into two groups of 30 patients each. The control group (R-group) received only Ropivacaine (150 mg of Ropivacaine 7.5% (20 ml) added to 2 ml of normal saline in the wound infiltration), while the intervention group (RD-group) received Ropivacaine with the addition of dexamethasone (150 mg of Ropivacaine 7.5% (20 ml) added to 8 mg of dexamethasone in the wound infiltration). Both groups were administered patient-controlled analgesia (PCA) with morphine for self-medication.

Postoperatively, a blinded evaluator assessed pain at H0, recorded the assessment of surgical scar pain using the Visual Analog Scale (VAS) at 4, 6, 12, 24, and 48 hours, as well as the time to the first opioid request, cumulative morphine consumption, opioid-related side effects, and length of stay. All patients were scheduled for a 3-month follow-up call to monitor chronic pain progression.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II and diagnosed with lumbar disc herniation, lumbar spinal stenosis, or lumbar degenerative spondylolisthesis requiring surgical treatment such as lumbar laminectomy and/or lumbar osteosynthesis.

Exclusion Criteria:

* Patients with altered communication capacity, previous spinal surgery, neuropathic pain, allergy to opioids, dexamethasone, or local anesthetics, active infection or tumor history, traumatic injury, chronic use of steroids or opioids, severe kidney, hepatic, or pulmonary failure, delayed extubation in post-anesthesia care unit (PACU), major bleeding during or after surgery, or surgical revision within the first 24 hours were excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-02-04 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
the time of the first analgesic demand of PCA | at 4, 6, 12, 24, and 48 hours postoperatively
  Change of VAS scores at 4, 6, 12, 24, and 48 hours postoperatively were also assessed by the patients after they had recovered from anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: ATEF BEN NSIR, PHD, Study Chair — HOPITAL UNIVERSITAIRE FATTOUMA BOURGUIBA
Locations (1):
- Hopital Fattouma Burguiba Monastir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No